CLINICAL TRIAL: NCT00733720
Title: Attenuation of Opioid Effects of Three Different Doses of Sublingual Buprenorphine / Naloxone by Oral Naltrexone in Healthy Volunteers
Brief Title: Buprenorphine Naltrexone-P1 A-Cocaine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Liza Gorgon, NIDA
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N01DA-6-8867
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2009-10

CONDITIONS: Cocaine-related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (1):
- 1 (Active Comparator): Each subject will receive all 3 doses of suboxone and placebo
  Interventions: Drug: Suboxone

INTERVENTIONS:
Drug: Suboxone — 4/1mg, 8/2mg 16/4mg
  Other Names: buprenorphine/naloxone; Subjects will be maintained on 50mg naltrexone

SUMMARY:
The purpose of this study is to determine if the opioid agonist effects of doses of 4/1 mg, 8/2 mg, and 16/4 mg of buprenorphine/naloxone can be completely blocked by 50 mg of oral naltrexone. This study will provide data to support the design of a similar study of the depot formulation of naltrexone and ultimately to study this combination for the treatment of cocaine dependence.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Be male/female between the ages of 18-55
* Be in good physical and mental health as determined by interview and physical exam
* Have a body mass index between 18 and 30, inclusive
* Have no oral cavity pathology that would interfere with sublingual absorption of buprenorphine/naloxone or placebo
* Have negative qualitative urine toxicology screen for opioids, cocaine, benzodiazepines, and barbiturates prior to administration of the first dose of naltrexone
* Be able to comply with protocol requirements
* If female, have a negative pregnancy test and agree to use an acceptable method of birth control from date of consent and until two weeks after the last administration of study drug or placebo

Exclusion Criteria:

* please contact site for more information

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Opioid Effects of study drug | daily

SECONDARY OUTCOMES:
Adverse Events | Daily

CONTACTS AND LOCATIONS:
Locations (1):
- Drug Dependence Research Center, San Francisco, California, United States